CLINICAL TRIAL: NCT05832489
Title: EEG-MRI Study of the Effect of Methylphenidate on Neural Mechanisms in Adult Patients With ADHD With or Without Mood Disorders: a Randomized Controlled Trial Versus Placebo
Brief Title: EEG-MRI Imaging of Methylphenidate Effects in Adult ADHD and Attentional Symptoms in Mood Disorders
Acronym: ImAteM-TDA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 7347
Record Dates: First submitted 2022-07-07; First posted 2023-04-27 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Adult ADHD; Adult-onset ADHD With Mood Disorder
Keywords: Adult ADHD; Sustained attention; fMRI; EEG; Pharmacoimaging; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Adult patients with ADHD (ADHD-P) receive a placebo or 25 mg of methylphenidate 45min before the first and second imaging sessions (MRI+EEG)
  Interventions: Drug: Placebo; Drug: Methylphenidate immediate release 25mg
- Group B (Experimental): Adult patients with attention deficit due to/emphasized by mood disorders (ADHD-HD) receive a placebo or 25 mg of methylphenidate 45min before the first and second imaging sessions (MRI+EEG)
  Interventions: Drug: Placebo; Drug: Methylphenidate immediate release 25mg
- Group C (Experimental): Adult Healthy controls receive a placebo or 25 mg of methylphenidate 45min before the first and second imaging sessions (MRI+EEG)
  Interventions: Drug: Placebo; Drug: Methylphenidate immediate release 25mg

INTERVENTIONS:
Drug: Placebo — Patients will have 2 imaging sessions (MRI and EEG) after either:
  * methylphenidate immediate release 25 mg
  * placebo
  in a cross-over design. The two imaging sessions will be separated by 11 to 87 days.
  Other Names: MRI; EEG
Drug: Methylphenidate immediate release 25mg — Patients will have 2 imaging sessions (MRI and EEG) after either:
  * methylphenidate immediate release 25 mg
  * placebo
  in a cross-over design. The two imaging sessions will be separated by 11 to 87 days.
  Other Names: MRI; EEG

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) in adults is a common psychiatric disorder, with important consequences in terms of quality of life, mental health (associated disorders and poorer response to treatment), family life, risk of accidents; with a consequent cost for society.

Adult ADHD is frequently associated with psychiatric co-morbidities, and notably associated with mood disorders (major depressive disorder or bipolar disorder) in about 50% of cases.

The diagnosis of ADHD in adults is made in patients with an attentional complaint (pure ADHD or ADHD-P), but also very often in the management of a comorbid mood disorder (ADHD associated with mood disorder, or ADHD-MD). In this case, the ADHD had no impact during childhood and adolescence.

Medication management is well established for ADHD-P, and medication is based on methylphenidate, which has a rapid and significant effect on attentional symptoms and impulsivity. However, in the case of ADHD-HD, there is little evidence of treatment efficacy and the mechanisms of action of methylphenidate at the brain level are poorly understood.

The aim of the study is to determine the neural mechanisms of the effect of methylphenidate, using functional MRI and EEG, in ADHD-P and ADHD-HD patients, and to compare them to healthy subjects. A single dose allows us to observe effects that are then persistent with repeated doses. The aim is to determine, by means of a biomarker, whether methylphenidate treatment responds to the same mechanisms in the different groups and would be relevant in ADHD-P as in ADHD-HD.

Main objective:

To determine whether methylphenidate impacts differently on brain circuits associated with cognitive functions in the two clinical populations studied (adult ADHD patients and patients with post mood disorder attentional deficit) and in comparison to controls.

Secondary objectives:

1. To determine the effect of methylphenidate on baseline brain flow in the two clinical populations and in controls (healthy subjects).
2. To determine whether methylphenidate has a different impact on cognitive performance in the two clinical populations studied and in comparison to controls (healthy subjects).
3. To confirm the effect of methylphenidate on the maintenance of cortical arousal.
4. To distinguish the brain networks impacted by methylphenidate (maintenance of attention or inhibition) with MRI and EEG.

DETAILED DESCRIPTION:
It is a cross-over, randomized, controlled, double-blind, study. 3 groups of 20 subjects are constituted: A: adult patients with ADHD (ADHD-P) B: patients with attention deficit due to/emphasized by mood disorders (ADHD-HD) C: healthy control population

During the inclusion visit the subjects fill in self-questionnaires (ASRS, WURS, WRAADDS, WFIRFS, TEMPS-A, BDI, BAI, RCTQ, mind-wandering). A 45-minute neuropsychological assessment will be carried out by a neuropsychologist, followed by training in the cognitive tasks used during the experimental sessions.

During imaging session 1 (3 to 60 days from inclusion):

Patients usually taking methylphenidate will discontinue methylphenidate treatment two days the imaging session.

Subject takes treatment (or placebo) 30-60 minutes before MRI. The MRI is performed at rest and associated with cognitive tasks (SART) (65 minutes duration). EEG is performed after in combination with a cognitive task (SART) (duration 40 minutes). Finally subjects complete self-questionnaires.

During imaging session 2 (14 to 90 days from inclusion): the same procedure is done again.

Patients usually taking methylphenidate will discontinue methylphenidate treatment two days before the session.

Subject takes placebo (if treatment during imaging session 1) or treatment (if placebo during imaging session 1) 30-60 minutes before MRI. MRI and EEG procedure are the same.

fMRI imaging includes rest and imaging during SART task (Go-NoGo), using BOLD and ASL sequences. EEG is performed during SART task.

ELIGIBILITY:
Inclusion criteria common to all groups:

* Subject (male or female) aged 18 to 60 years old
* Subject affiliated to a social protection health insurance scheme
* Subject capable of understanding the objectives and risks of the research and of providing dated and signed informed consent
* Subject having been informed of the results of the prior medical examination
* For a woman of childbearing age: negative blood pregnancy test and effective contraception throughout the study (intrauterine device, sterilization, estro-progestogen or progestogen per os, injectable or in the form of an implant or ring) and refusal to perform a pregnancy test before each MRI)

Inclusion criteria for Group A: ADHD patients without associated mood disorder (ADHD-P)

* Diagnosis of ADHD according to DSM-5 (in particular criterion B: presence of symptoms before the age of 12 years) NB: the diagnosis was not necessarily made at this age.
* Subject with or without methylphenidate treatment

Inclusion criteria for Group B: Patients with attention deficit disorder due to/accentuated by mood disorders (ADHD-MD)

* Association of ADHD symptoms with attentional disorders according to the combination of the following criteria :
* Diagnosis of Recurrent Depressive Disorder or Bipolar Disorder according to DSM-5
* Currently euthymic, i.e. a QIDS-16SC depression score < 6 and a YRMS mania score < 6, and clinically stabilized for at least 6 weeks prior to inclusion (stable and off-acute treatment). NB: for ISQ item 10 (concentration/decision making, score decision making only)
* DSM-5 Adult ADHD Criteria A (at least 5 symptoms of inattention and/or hyperactivity/impulsivity)
* Absence of Criterion D during childhood, adolescence and before mood disorders (i.e., no significant impact with reduced quality of social, academic or occupational functioning)
* Presence of Criterion D at present (symptoms have a significant impact with a reduction in the quality of social, academic or professional functioning)
* Subject with or without approved mood disorder treatment: Mood stabilizers (lithium, valproate, lamotrigine); antidepressants (SSRIs, IRSNa ≤60mg/j of venlafaxine and ≤60mg/j of duloxetine); benzodiazepines in stable doses for more than a month.
* Subject with or without methylphenidate treatment

Inclusion criteria for Group C: healthy subjects control

- Subject with no psychiatric or neurological history

Exclusion criteria common to all groups

* Subjects with contraindication to methylphenidate :

  * hypersensitivity to the active substance,
  * glaucoma,
  * pheochromocytoma,
  * treatment with other indirect sympathomimetics or alpha sympathomimetics (oral and/or nasal routes), irreversible MAOIs
  * Hyperthyroidism or thyrotoxicosis,
  * Pre-existing cardiovascular disorders including severe hypertension, heart failure, occlusive arterial disease, angina pectoris, congenital heart disease with hemodynamic impact, cardiomyopathy, myocardial infarction, arrhythmias and potentially life-threatening ductopathies (disorders caused by ion channel dysfunction),
  * Pre-existing cerebrovascular disorders, brain aneurysms, vascular abnormalities including vasculitis or stroke,
  * wheat allergy (other than celiac disease)
* Diagnosis or history of severe depression, anorexia nervosa or anorexic disorder, suicidal tendencies, psychotic symptoms, severe mood disorders, mania, schizophrenia, psychopathic or borderline personality disorder.
* Diagnosis or history of episodic and severe (type 1) (and poorly controlled) bipolar (affective) disorder.
* Subjectis with contraindication to performing an MRI: presence of non-removable ferromagnetic body, prosthesis, pacemaker, medication delivered by an implanted pump, vascular clip or stent, heart valve or ventricular shunt
* History that may affect brain anatomy or be related to an abnormality (neonatal suffering, neurosurgical operation, comitiality, stroke, head injury with unconsciousness of more than 15 minutes and mental retardation)
* History that may affect brain function (general anaesthesia or ECT within 3 months prior to inclusion)
* Substance Use Disorder as per DSM-5 criteria (except tobacco)
* Pregnant women or, in women of childbearing age and ability (non-sterile), lack of effective contraception
* Breastfeeding women
* Severe or unstable somatic pathology.
* Subject deprived of liberty, or in care under restraint
* Subject under safeguard of justice
* Incompetent subject (subject to a legal protection measure: curatorship, guardianship, future protection mandate, family habilitation)
* Impossibility to give informed information about the subject (subject in an emergency situation, difficulties in understanding the subject, ...)
* Subject in exclusion period defined by another protocol in progress

Exclusion criteria for Group A: ADHD patients without associated mood disorder (ADHD-P)

* Current Mood Disorder
* History of bipolar disorder in a first-degree relative
* Taking unauthorized psychotropic drugs: all antidepressants, antipsychotics, sedative antihistamines, regular hypnotics, benzodiazepines in unstable doses.

Exclusion criteria for Group B: Patients with attention deficit disorder due to/accentuated by mood disorders (ADHD-MD)

* Acute phase of mood disorder defined by scores a depression score in the QIDS-16SC ≥ 6 and a mania score in the YRMS ≥ 6. NB: for ISQ item 10 (concentration/decision making, score decision making only).
* Use of unauthorized psychotropic drugs including antipsychotics, sedative antihistamines, high-dose IRSNa (>150mg/d venlafaxine and >60mg/d duloxetine), MAOIs, tricyclic antidepressants, benzodiazepines in unstable doses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Effect of methylphenidate on the task vs. rest activation differential (treatment x group interaction) in a region defined by its involvement in the cognitive task and its responsiveness to methylphenidate. | 2 hours after intake of methylphenidate or placebo
  Changes in brain activations from J3-J600 to J14-J90 (MRI) in ADHD patients (ADHD-P and ADHD-HD), compared to healthy subjects(ADHD-P and ADHD-HD), compared to healthy subjects] ROI (Region of Interest) analysis to maximize power.

SECONDARY OUTCOMES:
Decrease in rCBF (regional Cerebral Blood Flow) in the methylphenidate vs. placebo condition, in the different groups (group x treatment interaction). | 2 hours after intake of methylphenidate or placebo
Improved cognitive performance in sustained attention and inhibition tasks (SART : number of errors) following methylphenidate administration, in the different groups. | 2 hours after intake of methylphenidate or placebo
EEG spectrum power in the low frequencies (proportion of delta power (1-4Hz) and theta power EEG bands (4-8Hz)) in the methylphenidate vs. placebo condition | 3 hours after intake of methylphenidate or placebo
MRI: Interaction group x treatment x task on brain activation related to sustained attention and inhibition corresponding to each of these tasks. | 2 hours after intake of methylphenidate or placebo
EEG evoked potentials: Interaction group x treatment x task on the amplitude of the P300 wave related to sustained attention (P300b) and related to inhibition (P300a) corresponding to each of these tasks. | 3 hours after intake of methylphenidate or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien WEIBEL, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Psychiatrie 2, Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No